CLINICAL TRIAL: NCT04661774
Title: Specific Effect of Foot Reflexology on Diaphragm Function: Comparison Between Different Biomarkers Upon Stimulation of the Reflex Area
Brief Title: Specific Effect of Foot Reflexology on Diaphragm Function
Acronym: FOOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: RC31/20/0251
Record Dates: First submitted 2020-11-06; First posted 2020-12-10 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Musculoskeletal Manipulations
Keywords: diaphragm dysfunction; reflexology
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: monocentric, interventional, comparative, randomized cross-over study in healthy individuals, with minimal risk and constraints
Who Masked: Participant
Masking Description: each participant has reflexology and placebo massage, he is his own comparator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham massage before reflexology massage (RP) (Other): Sham massage (MS) comparator will be realised before RP.
  Interventions: Other: reflexology massage; Other: sham massage
- Reflexology massage (RP) before Sham massage (Other): RP will be realized before Sham massage.
  Interventions: Other: reflexology massage; Other: sham massage

INTERVENTIONS:
Other: reflexology massage — reflexology massage of the foot zone implicated in diaphragm stimulation
Other: sham massage — traditional massage of the foot

SUMMARY:
Diaphragm dysfunction, are refractory to drug therapy. This encourage investigators to explore new non-drug therapeutic paths, such as plantar reflexology (RP). The investigators proposed a comparison of the evolution of different parameters, quantitative and qualitative, to identify biomarkers and highlight the specific effect of RP on the diaphragm function, compared to placebo.

DETAILED DESCRIPTION:
Many complex, chronic and multifactorial dysfunctions, such as diaphragm dysfunction, are refractory to drug therapy. This encourage investigators to explore new non-drug therapeutic paths, such as plantar reflexology (RP). This change is essential and will broaden relevant solutions to health.

Despite the very positive benefits of RP highlighted, the methodological quality of trials are often poor and there are gaps notably on the description of the intervention, the blind, the drop-out rate ... which prevents the meta-analyzes to conclude. Promoting rigorous research will play an essential role in the transition to personalized and integrative medicine. With the intention of specifying the methods of application and the indications of the PR, it is necessary to correctly evaluate and be able to cross-check the different information It therefore seems relevant to combine research on the objective physiological effects in correlation with the patient's subjective feelings to initiate the scientific validation of RP and thus non-drug interventions as recommended by the High Authority for Health (HAS). The hypothesis is that through a comparison of the evolution of different parameters, quantitative and qualitative, this study will allow to identify biomarkers and highlight the specific effect of RP on the diaphragm function, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 20 to 40
* Healthy right-handed subject, attested by a score ≥ 8/10 on the Edinburgh manual laterality questionnaire
* Naive subject in Reflexology.

Exclusion Criteria:

* Contraindication to carrying out the MRI examination
* Subject refusing to be informed of any abnormality detected on brain MRI,
* Subject presenting a neurodegenerative disease,
* Subject presenting a cardiac disease,
* Subject presenting skin lesions in the feet or recent fracture in the feet,
* Subject having an history of phlebitis less than 3 months
* Subject having an history of deep vein thrombosis.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
modulation of brain activity of the specific impact of RP | day 1
  a comparison between the activation cards of the brain networks and a map of correlation coefficients representing the strength of the connectivity between the different brain networks and regions of interest

SECONDARY OUTCOMES:
variation of physiological constants related to the function of the diaphragm | Day 1
  collection of respiratory rate
variation of physiological constants related to the function of the diaphragm | Day 1
  collection of saturation
variation in physiological constants linked to the ANS | Day 1
  collection of heart rate
subjective feelings of the subjects | Day 1
  Likert scale for the subjective assessment of stress and a Likert scale for the subjective assessment of ease of breathing (graduations from 1 to 7 with 1 = I completely agree and 7= I Don't agree at all)

CONTACTS AND LOCATIONS:
Locations (1):
- PAYOUX, Toulouse, France

IPD SHARING:
Plan to Share IPD: No